CLINICAL TRIAL: NCT06151080
Title: An Open, Single-arm Clinical Study of Lenalidomide Combined With G-CHOP(LO-CHOP) in the Treatment of Newly Diagnosed Diffuse Large B-cell Lymphoma With Follicular Lymphoma (CDLBCL-FL).
Brief Title: Lenalidomide Combined With G-CHOP in the Treatment of Newly Diagnosed DLBCL With FL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Sun Yat-sen University (Other); Jiangxi Provincial Cancer Hospital (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-01
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LO-CHOP (Experimental): Lenalidomide combined with G-CHOP
  Interventions: Drug: Lenalidomide combined with G-CHOP (LO CHOP)

INTERVENTIONS:
Drug: Lenalidomide combined with G-CHOP (LO CHOP) — Lenalidomide combined with G-CHOP to treat newly diagnosed diffuse large B-cell lymphoma with follicular lymphoma (CDLBCL-FL)

SUMMARY:
To evaluate the efficacy and adverse effects of lenalidomide combined with G-CHOP(LO-CHOP) in the treatment of newly diagnosed diffuse large B-cell lymphoma with follicular lymphoma (CDLBCL-FL).

DETAILED DESCRIPTION:
This is a Phase 2, open-label clinical trial study that aims to evaluate the efficacy (Complete response, Overall Survival, Progression Free Survival) and adverse effects of lenalidomide combined with G-CHOP(LO-CHOP) in the treatment of newly diagnosed diffuse large B-cell lymphoma with follicular lymphoma (CDLBCL-FL).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old, gender is not limited;
2. According to the REAL/WHO classification, the newly diagnosed diffuse large b-cell lymphoma with follicular lymphoma (CDLBCL-FL): the same lymph node specimen showed diffuse large b-cell lymphoma and follicular lymphoma, or the tissue specimen showed diffuse large b-cell lymphoma and indolent lymphoma in bone marrow pathology; or the different group specimens suggested diffuse large b-cell lymphoma and/or follicular lymphoma, respectively, with stage II-IV.
3. Using the Lugano 2014 lymphoma response evaluation criteria, there must be at least one measurable or evaluable lesion: PET/CT can evaluate the lesion, CT or MRI can evaluate the lesion in the node with a diameter greater than 1.5 cm, a short diameter greater than 1.0 cm, or an extranodal lesion with a diameter greater than or equal to 1.0 cm
4. ECOG 0-2
5. Left ventricular ejection fraction (LVEF) was less than 45%
6. HBV-positive serology (occult carriers: anti-HBeAg +, anti-HBsAg-, anti-HBsAg +/-) can only be enrolled if the HBV-dna test is negative.
7. Normal major organ function: liver function: serum bilirubin ≤2.0 × ULN, serum ALT and AST ≤2.5 × ULN, renal function: serum CR ≤2.0 × ULN; (unless caused by lymphoma)
8. Absolute neutrophil count (ANC)≥1.0 × 109 l, platelet count (PLT)≥100 × 109 L, hemoglobin content (HGB)≥80 g L, if myeloma was involved, ANC ≥0.75 × 109 L, platelet count (PLT)≥50 × 109 L, HGB content (HGB) was not required.
9. Life expectancy ≥6 months
10. Informed consent (all studies had to sign a patient's informed consent form)

Exclusion Criteria:

1. DLBCL of primary and secondary centers;
2. HIV-positive patients and/or HCV-active infections (recorded through HCV-RNA-positive testing)
3. Clinically evident secondary cardiovascular diseases such as uncontrollable hypertension (resting diastolic pressure>115 mmHG), uncontrolled arrhythmias, symptomatic angina pectoris, or NYHA III-IV congestive heart failure.
4. Severe chronic obstructive pulmonary disease complicated with hypoxemia.
5. Active bacterial, fungal, and/or viral infections beyond the control of systemic therapy
6. Except for cured skin basal cell carcinoma or cervical carcinoma in situ, or early prostate cancer that does not require systemic treatment or early breast cancer only requires surgery. Other malignant tumors have occurred within the past 3 years or at the same time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | Up to 28 months
  Complete remission rate was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Progression-free survival | From the randomization until the first documentation of PD or death whichever occurs first or up to 28 months
  PFS was defined as the time from the date of treatment initiation to the date of first documentation of definitive disease progression (PD) or date of death from any cause, whichever occurs first.
Overall survival | Up to 28 months
  OS will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, PhD, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No